CLINICAL TRIAL: NCT05151692
Title: A Sequential, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of JNJ-80202135 Following a Single Intravenous Administration in Healthy Chinese Adult Participants
Brief Title: A Study of JNJ-80202135 in Healthy Chinese Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CR109100; 80202135EDI1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-12-07; First posted 2021-12-09 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1: Nipocalimab (Experimental): Participants will receive a single intravenous (IV) dose of nipocalimab Dose 1 on Day 1.
  Interventions: Drug: Nipocalimab
- Cohort 2: Nipocalimab (Experimental): Participants will receive a single IV dose of nipocalimab Dose 2 on Day 1.
  Interventions: Drug: Nipocalimab
- Cohort 3: Nipocalimab (Experimental): Participants will receive a single IV dose of nipocalimab Dose 3 on Day 1.
  Interventions: Drug: Nipocalimab

INTERVENTIONS:
Drug: Nipocalimab — Nipocalimab will be administered as an IV infusion.
  Other Names: JNJ-80202135

SUMMARY:
The purpose of this study is to assess the pharmacokinetic (PK) of nipocalimab following single intravenous (IV) administration in healthy Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, vital signs and 12-lead electrocardiogram (ECG) performed at screening. If there are any abnormalities, they must be assessed as not clinically significant by the investigator and this determination must be recorded in the participant's source documents and initialed by the investigator
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Serum immunoglobulin G (IgG) level must be greater than (>) the lower limit of normal at screening
* Body mass index (BMI; weight [kilograms {kg}] per height^2 [meter square {m^2}]) between 18 and 27.9 kilograms per meter square (kg/m^2) (inclusive), and body weight not less than 50 kg and less than or equal to (<=) 110 kg at screening
* A woman of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at Week 0 prior to administration of study intervention

Exclusion Criteria:

* Known allergies, hypersensitivity, or intolerance to nipocalimab or its excipients
* Serum albumin below the lower limit of normal at screening
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol, acetaminophen, contraceptives, and hormonal replacement therapy within 14 days before the first dose of the study drug is scheduled until completion of the study
* Had major surgery, (example: requiring general anesthesia) within 12 weeks before screening, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study or within 8 weeks after the last dose of study intervention administration
* Has an active, acute or a chronic infection (examples: bronchiectasis, chronic osteomyelitis, chronic pyelonephritis) or requires chronic treatment with anti-infectives (examples: antibiotics, antivirals)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Area Under the Serum Concentration Versus Time Curve From Time Zero to Time of the Last Measurable Concentration (AUC[0-last]) of Nipocalimab | Up to Day 29
  AUC(0-last) is defined as area under the serum concentration versus time curve from time 0 to time of the last measurable concentration of nipocalimab.
Area Under the Analyte Concentration Versus Time Curve From Time Zero to Infinite Time (AUC [0-Infinity]) of Nipocalimab | Up to Day 29
  AUC (0-Infinity) is defined as area under the analyte concentration versus time curve from time zero to infinite time of nipocalimab.
Last Measurable Serum Concentration (Clast) of Nipocalimab | Up to Day 29
  Clast is defined as last measurable serum concentration of nipocalimab.
Maximum Observed Serum Concentration (Cmax) of Nipocalimab | Up to Day 29
  Cmax is defined as maximum observed serum concentration of nipocalimab.
Time of Last Measurable Serum Concentration (Tlast) of Nipocalimab | Up To Day 29
  Tlast is defined as time of last measurable serum concentration of nipocalimab.
Time to Reach the Maximum Observed Serum Concentration (Tmax) of Nipocalimab | Up to Day 29
  Tmax is defined as time to reach the maximum observed serum concentration of nipocalimab.
Apparent Elimination Half-life (T1/2) of Nipocalimab | Up to Day 29
  T1/2 is defined as apparent elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve of nipocalimab.
Total Systemic Clearance (CL) of Nipocalimab | Up to Day 29
  CL is defined as total systemic clearance of nipocalimab after intravenous (IV) administration.
Volume of Distribution (Vz) of Nipocalimab | Up to Day 29
  Vz is defined as volume of distribution based on terminal phase after IV administration of nipocalimab.

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to Day 57
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study.
Percentage of Participants with Serious Adverse Event (SAE) | Up to Day 57
  A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Percentage of Participants with Adverse Event of Special Interests (AESIs) | Up to Day 57
  Percentage of participants with AESIs will be reported. Treatment-emergent AEs associated with the following situations are considered as AESI: a) severe or medically significant or immediately life-threatening infections requiring IV anti-infective or operative/invasive intervention or requiring hospitalization or prolongation of existing hospitalization; b) hypoalbuminemia with albumin less than (<) 20 grams per liter (g/L). Any AE occurring at or after the initial administration of study intervention through end of study is considered to be treatment-emergent.
Percentage of Participants with Abnormalities in Physical Examinations | Up to Day 57
  Percentage of participants with abnormalities in physical examinations (including height and body weight) will be reported.
Percentage of Participants with Abnormalities in 12-Lead Electrocardiogram (ECG) Values | Up to Day 57
  Percentage of participants with abnormalities in 12-lead ECG values will be reported.
Percentage of Participants with Abnormalities in Vital Signs | Up to Day 57
  Percentage of participants with abnormalities in vital signs (temperature axillary, pulse/heart rate, blood pressure [systolic and diastolic]) will be reported.
Percentage of Participants with Abnormalities in Clinical Laboratory Values | Up to Day 57
  Percentage of participants with abnormalities in clinical laboratory values (hematology, clinical chemistry, urinalysis) will be reported.
Percentage of Participants with Anti-drug Antibodies to Nipocalimab | Day 1, Day 15, Day 29 and Day 57
  Percentage of participants with anti-drug antibodies to nipocalimab will be reported.
Change from Baseline Over Time in Total Immunoglobulin-G (IgG) Serum Levels | Baseline up to Day 57
  Change from baseline over time in total IgG serum levels will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Li H, Liu J, Wang X, Zhao W, Zhang L, Niu X, Liu J, Dong Z. Pharmacokinetics, Pharmacodynamics, and Safety of Nipocalimab in Healthy Chinese Volunteers: A Single-Dose, Phase I Study. Neurol Ther. 2025 Aug;14(4):1439-1450. doi: 10.1007/s40120-025-00763-5. Epub 2025 May 19. PMID 40389701